CLINICAL TRIAL: NCT04765748
Title: Cytokine Filter Usage During Open Thoracoabdominal Aortic Aneurysm Repair- a Single-center Randomized Prospective Trial- Cytosorb and Its Imapct on Open TAAA Repair Outcome
Brief Title: Cytokine Filter Usage During Open Thoracoabdominal Aortic Aneurysm Repair- a Single-center Randomized Prospective Trial
Acronym: TAAA-Cytosorb
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Alexander Gombert, Principle Investigator PD Dr. med. Alexander Gombert, Specialist in Vascular Surgery, RWTH Aachen University
Other Study IDs: 20-031
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Complications; Inflammatory Response
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAAA patients with Cytosorb: Patients suffering from a TAAA larger than 55mm
  Interventions: Device: Cytosorb
- TAAA patients without Cytosorb: Patients suffering from a TAAA larger than 55mm

INTERVENTIONS:
Device: Cytosorb — Cytokine filter, which can be used intraoperatively while using a heart lung machine
  Groups: TAAA patients with Cytosorb

SUMMARY:
Prospecrtive study including 20-30 randomized patients treated by open repair because of an TAAA larger than 55 mm During the surgery, a heart lung machine is applied for distal perfusion during aortic cross clamping to enable distal organ perfusion.

Regardless an intensive inflammatory reaction is a well known effect after reperfusion, leading to a uncontrolled inflammation during th first days after surgery. This may be associated to bad outcome and decreased survival rates. By the application of a intraoperative cytokine and DAMP filter this negative ffect could be reduced, resulting in a better outcome after surgery.

DETAILED DESCRIPTION:
Prospecrtive study including 20-30 randomized patients treated by open repair because of an TAAA larger than 55 mm During the surgery, a heart lung machine is applied for distal perfusion during aortic cross clamping to enable distal organ perfusion.

Regardless an intensive inflammatory reaction is a well known effect after reperfusion, leading to a uncontrolled inflammation during th first days after surgery. This may be associated to bad outcome and decreased survival rates. By the application of a intraoperative cytokine and DAMP filter this negative ffect could be reduced, resulting in a better outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

Suffering from a TAAA larger than 55mm

Exclusion Criteria:

immunosupprive therapy pregnancy

-

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients treated by open TAAA repair
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Amount of perioperative catecholamine usage in mg/dl for the first seven days after surgery | 7 days perioperatively -10 day postoperatively
  amount measured in mg/dl
Amount of transfusion required during and after the surgery, assessed in transfusion more or less than 5 blood bags | 7 days perioperatively 5-10 day postoperatively
  packed cells, erythrocyte concentrate

SECONDARY OUTCOMES:
Acute kidney injury, measured using serum creatinine in mg/dl | 7 days perioperatively, -10 day postoperatively
  AKI assessed according to the KDIGO classification perioperatively for the first 7 days after surgery
Patients survival for the first 12 months after surgery | 12 months 10-14 months postopertaibely
  Survival yes/no within the first 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Alexander Gombert, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No